CLINICAL TRIAL: NCT07241806
Title: Correlation Between Axial Length and Degree of Refractive Error With Optic Disc Parameters , Ganglion Cell Complex and Peripapillary RNFL Thickness
Brief Title: Measurment of Optic Disc Parameters, RNFL Thickness and Ganglion Cell Complex in Myopic, Hypermetropic and Emmetropic Patients Using OCT and Axial Length Measurments
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariam Smeh Roshdy, doctor, Assiut University
Other Study IDs: OCT in refractive error
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Refractive Errors
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: OCT — Axial length measurement (using A-scan)
  Spectral-domain OCT: All the patients will undergo OCT imaging using NIDEK RS-330 Retina scan duo 2 (SD-OCT)(CO-LTD made in Japan 2017) with scan speed 70.000 axial scans per second and wavelength of 880 nm for:
  Peripapillary RNFL thickness in all quadrants GCC thickness (average, superior, inferior,nasal,temporal) Optic disc parameters (disc area, cup/disc ratio, rim area)

SUMMARY:
To evaluate the optic disc parameters, thickness of ganglion cell complex (GCC), and thickness of peripapillary retinal nerve fiber layer (RNFL) in myopic and hyperopic and emmetrop patients using optical coherence tomography (OCT), and to correlate these changes with axial length and degree of refractive error.

DETAILED DESCRIPTION:
Refractive errors, particularly myopia and hyperopia, are among the most common ocular conditions globally, affecting both children and adults .

Myopia is frequently associated with axial elongation, which may induce structural changes in the posterior segment of the eye such as thinning of the peripapillary retinal nerve fiber layer (RNFL) and alteration of optic disc parameters . Hyperopia, conversely, is linked to shorter axial lengths and has been shown to affect retinal and optic nerve anatomy in distinct ways .

Optical coherence tomography (OCT), particularly spectral-domain OCT (SD-OCT), allows for high-resolution imaging of the RNFL and ganglion cell complex (GCC), which are crucial for visual processing. These layers are known to undergo subtle changes not only due to disease processes like glaucoma or optic neuropathies but also as a result of anatomical differences induced by refractive status .

While many studies have independently evaluated RNFL or GCC in myopic and hyperopic patients, few have directly compared these two refractive states while correlating structural findings with axial length and refractive error magnitude . Including an emmetropic control group provides a normative benchmark, enhancing the clinical relevance of the findings .

This study seeks to fill this gap by offering a comparative structural analysis using OCT, aiming to enhance diagnostic sensitivity and understanding of optic nerve and macular changes in various refractive profiles.

ELIGIBILITY:
Inclusion Criteria:

* Adults age starting from 18 years old Diagnosed with myopia (≤ -0.50 D) or hyperopia (≥ +0.50 D) Clear ocular media for high-quality OCT imaging No prior ocular surgeries Willing to provide informed consent IOP below 21

Exclusion Criteria:

* Presence of glaucoma or optic nerve pathologies Retinal diseases or degenerative changes Systemic diseases affecting the eye (e.g., diabetes, hypertension) History of trauma or intraocular surgery High astigmatism (> ±2.00 D) Poor OCT image quality

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults age starting from 18 years old Diagnosed with myopia (≤ -0.50 D) or hyperopia (≥ +0.50 D) Clear ocular media for high-quality OCT imaging No prior ocular surgeries Willing to provide informed consent IOP below 21 exculuding Presence of glaucoma or optic nerve pathologies Retinal diseases or degenerative changes Systemic diseases affecting the eye (e.g., diabetes, hypertension) History of trauma or intraocular surgery High astigmatism (> ±2.00 D) Poor OCT image quality
Sampling Method: Non-Probability Sample
Enrollment: 266 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the optic disc parameters, thickness of ganglion cell complex (GCC), and thickness of peripapillary retinal nerve fiber layer (RNFL) in myopic and hyperopic and emmetrop patients using optical coherence tomography (OCT) | two years
  To evaluate the optic disc parameters, thickness of ganglion cell complex (GCC), and thickness of peripapillary retinal nerve fiber layer (RNFL) in myopic and hyperopic and emmetrop patients using optical coherence tomography (OCT)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Holden BA, Fricke TR, Wilson DA, Jong M, Naidoo KS, Sankaridurg P, Wong TY, Naduvilath TJ, Resnikoff S. Global Prevalence of Myopia and High Myopia and Temporal Trends from 2000 through 2050. Ophthalmology. 2016 May;123(5):1036-42. doi: 10.1016/j.ophtha.2016.01.006. Epub 2016 Feb 11. PMID 26875007
- [Result] Chen Y, Li X, Wang J, et al. Recent large-sample findings reinforcing the relationship between myopia (axial elongation) and reduced RNFL thickness, with discussion of magnification correction. Sci Rep. 2024;14(1):12567.
- [Result] Wu Z, Huang J, Wang Y, et al. Retinal structural changes associated with high refractive errors: A comparative OCT analysis. Eye (Lond). 2024;38(1):112-120.
- [Result] Hougaard JL, Wang M, Fjeldstad JS. Quantitative OCT findings in high myopia and hyperopia. Acta Ophthalmol. 2023;101(4):e315-e322.
- [Result] Liu S, Chen J, Xu Y, Li Y, Zhang X. Effects of refractive error on GCC and RNFL thickness: a meta-analysis. Eye Vis (Lond). 2023;10(1):14
- [Result] Wang D, Zhang Y, Chen H, Li L, Zhou Y. Evaluation of RNFL thickness in hyperopic eyes: a comparative OCT-based study. Int J Ophthalmol. 2022;15(4):599-605.
- [Result] . Leung CK, Yu M, Weinreb RN, Mak HK, Lai G, Ye C, et al. Impact of axial length on optic disc and retinal nerve fiber layer measurements. Invest Ophthalmol Vis Sci. 2011;52(1):291-9.
- [Result] . Kim M, Choi EH, Lee HS, Park SW, Kim JH, Yu YS. Peripapillary and macular retinal thickness in high myopia measured with OCT. BMC Ophthalmol. 2020;20(1):285.
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/26875007/